CLINICAL TRIAL: NCT00599248
Title: A Phase 1 Study to Determine the Safety and Biological Activity of Cell-Mediated Gene Therapy Using TissueGene-C in Patients With Degenerative Joint Disease Prior to Total Knee Arthroplasty
Brief Title: Safety Study of TissueGene-C in Degenerative Joint Disease of the Knee
Acronym: TGC-03-01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kolon TissueGene, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TGC-03-01
Record Dates: First submitted 2008-01-11; First posted 2008-01-23 (Estimated); Results first posted 2016-06-30 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-06

CONDITIONS: Osteoarthritis, Knee
Keywords: osteoarthritis, knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): TissueGene-C single intraarticular injection of 3x10e6 cells/joint
  Interventions: Biological: TissueGene-C
- 2 (Experimental): TissueGene-C single intraarticular injection of 1x10e7 cells/joint
  Interventions: Biological: TissueGene-C
- 3 (Experimental): TissueGene-C single intraarticular injection of 3x10e7 cells/joint
  Interventions: Biological: TissueGene-C
- 4 (Placebo Comparator): Placebo control single intraarticular injection
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: TissueGene-C — TissueGene-C at 3x10e6, 1x10e7 or 3x10e7 cells/joint to be administered by intra-articular injection
  Arms: 1; 2; 3
Biological: Placebo — Placebo control (DMEM)
  Arms: 4

SUMMARY:
The study is being conducted to investigate the safety and activity of TissueGene-C injected into the knee joint of patients with chronic degenerative joint disease (DJD) who will be undergoing total knee replacement.

DETAILED DESCRIPTION:
The purpose of this first human study is to investigate the safety and biological activity of intra-articularly applied TissueGene-C in patients with chronic degenerative joint disease (DJD) who will be undergoing total knee replacement. In addition, data on joint pain, range of motion, and functionality will be obtained in this patient population prior to total knee replacement.

The primary objective of this study is to evaluate the safety and biological activity of intra-articularly administered TissueGene-C as evidenced by observation of the injection site for irritation or other abnormalities affecting the incidence and severity of adverse events, and the changes in physical examination findings and laboratory tests as compared to the placebo control.

The secondary objectives of this study are to:

1. Evaluate the dose response of the hChonJb#7 cells in grafting at the defect as compared to the placebo control.
2. Evaluate distribution of hChonJb#7 cells out of the injection site.
3. Evaluate the regeneration of hyaline cartilage as determined by the histological analysis of the resected knee tissue.
4. Evaluate the joint for evidence of tissue overgrowth or transformation.
5. Evaluate the biological activity of TissueGene-C on joint pain, range of motion and functionality as compared to the placebo control

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female subjects
2. Age 18 years and older
3. In general good health as evidenced by physical examination, normal hematology, serum chemistry, and urinalysis screening laboratory results, and a negative history of significant organ system disorders. All laboratory values must be within 20% of normal ranges.
4. Patients with Degenerative Joint Disease (DJD) of the knee that is refractory to existing drug therapies and who are scheduled for Total Knee Arthroplasty.
5. Based on Radiographic findings, defect should be more than 2 cm.
6. Patients providing written informed consent, after the nature of the study, are fully explained.
7. Body Mass Index (BMI) should be between '18.5 - 45.5'. The applied scale is the same for both men and women.
8. Blood Pressure measurements - Systolic Blood Pressure (SBP) should be between 90-160mm. Hg, and Diastolic Blood Pressure (DBP) between 50-90mm.Hg,
9. Osteoarthritis confirmed by the Radiographic Criteria of Kellgren and Lawrence
10. Symptom of pain for more than four (4) consecutive months and intensity greater than Grade 4 on the 11-point numeric scale.

Exclusion Criteria:

1. Patients with abnormal hematology, serum chemistry, or urinalysis screening laboratory results
2. Patients taking anti-inflammatory medications (prescription or over-the-counter), including herbal therapies, within 14 days of baseline visit
3. Patients with a recent (within 1 year) history of drug abuse and/or a positive urine drug/alcohol test at the time of screening
4. Patients receiving injections to the treated knee within 2 months prior to study entry
5. Patients who are pregnant or currently breast-feeding children
6. Patients with systemic, rheumatic, or inflammatory disease of the knee or chondrocalcinosis, hemochromatosis, inflammatory arthritis, necrosis of the femoral condyle, arthropathy of the knee associated with juxta-articular Paget's disease of the femur or tibia, ochronosis, hemophilic arthropathy, infectious arthritis, Charcot's knee joint, villonodular synovitis, and synovial chondromatosis.
7. Patients with ongoing infectious disease, including HIV and hepatitis
8. Patients with clinically significant cardiovascular, renal, hepatic, endocrine disease, cancer, or Type I diabetes
9. Patients participating in a study of an experimental drug or medical device within 30 days of study entry.
10. Positive drug screen at screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-01; Primary Completion 2009-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mont, MD, Principal Investigator — Sinai Hospital of Baltimore; David Romness, MD, Principal Investigator — Commonwealth Orthopedics, Virginia Hospital Center
Locations (2):
- United States (2):
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Commonwealth Orthopedics, Arlington, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment and assignment of patients in Arms 2 and 3 (dose escalation to sequentially higher doses) was only performed after completion of review of safety data in the previous Arm (lower dose) by the Independent Data Monitoring Committee
Groups:
- Active Treatment (TG-C) 1: TissueGene-C at 3x10e6 cells/joint
  TissueGene-C: TissueGene-C at 3x10e6 cells/joint administered by single intra-articular injection
- Active Treatment (TG-C) 2: TissueGene-C at 1 x 10e7 cells/joint
  TissueGene-C: TissueGene-C at 1x10e7 cells/joint administered by single intra-articular injection
- Active Treatment (TG-C) 3: TissueGene-C at 3x10e7 cells/joint
  TissueGene-C: TissueGene-C at 3x10e7 cells/joint administered by single intra-articular injection
- Placebo Control (DMEM): Placebo Control (DMEM)
  Placebo: Placebo control (DMEM) administered by a single intraarticular injection
Period: Overall Study
Arm/Group | Active Treatment (TG-C) 1 | Active Treatment (TG-C) 2 | Active Treatment (TG-C) 3 | Placebo Control (DMEM)
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Adults 18 or older with degenerative joint disease of the knee (confirmed by Kellgren and Lawrence criteria) refractory to existing drug therapies who were scheduled for total knee arthroplasty.
Groups:
- Active Treatment (TG-C): TissueGene-C at 3x10e6, 1x10e7 or, 3x10e7 cells/joint
  TissueGene-C: TissueGene-C at 3x10e6, 1x10e7 or 3x10e7 cells/joint to be administered by intra-articular injection
- Placebo Control (DMEM): Placebo control
  Placebo: Placebo control (DMEM)
- Total: Total of all reporting groups
Arm/Group | Active Treatment (TG-C) | Placebo Control (DMEM) | Total
Number analyzed (Participants) | 9 | 3 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 3 | 10
  >=65 years | 2 | 0 | 2
Age, Continuous [Median (Full Range); unit: Years] | 61.0 [39 to 67] | 60.0 [36 to 61] | 60.5 [36 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 2 | 10
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 9 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Summary of Adverse Events
Description: The incidence of observations at the site of administration and the incidence adverse events assessed through 28 days after treatment.
Time Frame: Through 28 days post-dosing
Population: Intention-to-treat
Measure: Number; unit: Adverse events
Groups:
- Active Treatment (TG-C) 1: TissueGene-C at 3x10e6 cells/joint
  TissueGene-C: TissueGene-C at 3x10e6 cells/joint to be administered by a single intra-articular injection
- Active Treatment (TG-C) 2: TissueGene-C at 1x10e7 cells/joint
  TissueGene-C: TissueGene-C at 1x107 cells/joint to be administered by a single intra-articular injection
- Active Treatment (TG-C) 3: TissueGene-C at 3x10e7 cells/joint
  TissueGene-C: TissueGene-C at 3x10e7 cells/joint to be administered by a single intra-articular injection
Arm/Group | Active Treatment (TG-C) 1 | Active Treatment (TG-C) 2 | Active Treatment (TG-C) 3 | Placebo Control (DMEM)
Number analyzed (Participants) | 3 | 3 | 3 | 3
Adverse events | 2 | 2 | 3 | 2

2. Secondary Outcome: Number of Patients Showing Engraftment at the Defect
Description: Dose Response of the TG-C in Engrafting at the Defect as Compared to Placebo Control
Time Frame: 28 Days
Measure: Number; unit: participants
Groups:
- Active Treatment (TG-C) 2: TissueGene-C at 1x10e7 cells/joint
  TissueGene-C: TissueGene-C at 1x10e7 cells/joint to be administered by a single intra-articular injection
Arm/Group | Active Treatment (TG-C) 1 | Active Treatment (TG-C) 2 | Active Treatment (TG-C) 3 | Placebo Control (DMEM)
Number analyzed (Participants) | 3 | 3 | 3 | 3
participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Patients With Distribution of hChonJb#7 Cells Detected Outside of the Injection Site
Description: Number of Patients with Distribution of hChonJb#7 Cells Detected Outside of the Injection Site as determined by PCR analysis for vector DNA.
Time Frame: 12 Months
Measure: Number; unit: participants
Arm/Group | Active Treatment (TG-C) 1 | Active Treatment (TG-C) 2 | Active Treatment (TG-C) 3 | Placebo Control (DMEM)
Number analyzed (Participants) | 3 | 3 | 3 | 3
participants | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Observable Evidence of Cartilage Regeneration
Description: The evaluation of regeneration of hyaline cartilage as determined by histological analysis of resected knee tissue and observation for engraftment and cartilage production.
Time Frame: Days 0, 3, 7, 11, 28 (prior to surgery), and day 29 (one day post-surgery) following dosing. Follow-up patient monitoring will be performed at 3, 6, 9, and 12 months following dosing
Population: Intention-to-treat
Measure: Number; unit: participants
Arm/Group | Active Treatment (TG-C) 1 | Active Treatment (TG-C) 2 | Active Treatment (TG-C) 3 | Placebo Control (DMEM)
Number analyzed (Participants) | 3 | 3 | 3 | 3
participants | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Patients With Tissue Overgrowth or Transformation in the Knee Joint
Description: Visual and histological analysis of knee joint tissues to determine the number of patients with tissue overgrowth or transformation
Time Frame: 29
Measure: Number; unit: participants
Arm/Group | Active Treatment (TG-C) 1 | Active Treatment (TG-C) 2 | Active Treatment (TG-C) 3 | Placebo Control (DMEM)
Number analyzed (Participants) | 3 | 3 | 3 | 3
participants | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Patients With Improvements in Pain and Function of the Knee Joint
Description: Assessment of the number of patients with improvement in pain and function of the knee joint
Time Frame: 28 Days
Measure: Number; unit: participants
Arm/Group | Active Treatment (TG-C) 1 | Active Treatment (TG-C) 2 | Active Treatment (TG-C) 3 | Placebo Control (DMEM)
Number analyzed (Participants) | 3 | 3 | 3 | 3
participants | 3 | 3 | 3 | 3

ADVERSE EVENTS:
Time Frame: 1 Year
Description: Treatment emergent adverse events
Arm/Group | Active Treatment (TG-C) | Placebo Control (DMEM)
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/3
Other Adverse Events (participants affected / at risk) | 7/9 | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Treatment (TG-C) (N=9) | Placebo Control (DMEM) (N=3)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lower extremity mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Activated PTT prolonged (Investigations) | 2 (2) | 1 (1)
PT Prolonged (Investigations) | 1 (1) | 1 (1)
Blood test abnormal (Investigations) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (1)
Pruritis generalized (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Rhinitis allgergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was designed a a preliminary assessment of safety in a limited population (12 subjects: 9 active 3 placebo) therefore statistics are presented descriptively.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days